CLINICAL TRIAL: NCT07389512
Title: Development and Evaluation of Clinical Radiopharmacy in the Pharmaceutical Management of Patients Treated With Targeted Radionuclide Therapy (TRT) Within Nuclear Medicine Departments
Brief Title: Pharmaceutical Management in Targeted Radioligand Therapy
Acronym: PharmTRT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0917; 25-5201 (Other: HCL)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Thyroid Cancer; Metastatic Prostate Cancer; Neuroendocrine Tumor Carcinoid
Keywords: Clinical radiopharmacy; Pharmaceutical consultation; Targeted Radionuclide Therapy
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms; Prostatic Neoplasms; Carcinoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TRT Cohort: Cohorte of patients treated with Targeted Radionuclide Therapy for thyroid cancer

SUMMARY:
Targeted Radionuclide Therapy (TRT) is a treatment modality used in nuclear medicine to target cancer cells while preserving surrounding healthy tissues. This approach is based on the use of radiopharmaceuticals (RPs)-compounds that combine a radioactive isotope with a molecule designed to selectively bind to cancer cells.

TRT has historical roots, dating back to the 1950s with the introduction of radioactive iodine-131. It has long been used for the treatment of thyroid cancers, which require hospitalization for 3 to 5 days in a dedicated, isolated, and radioprotected environment.

In recent years, TRT has undergone significant development with the emergence of new isotopes coupled with innovative molecules targeting a wider range of cancers. Lutathera ([177Lu]Lu-DOTATATE) and Pluvicto ([177Lu]Lu-PSMA-617), available since 2021, have revolutionized the management of patients with neuroendocrine tumors and metastatic prostate cancer, respectively. Numerous clinical trials are currently underway or planned, further expanding the field. These cutting-edge treatments are administered intravenously-mostly on an outpatient basis-within nuclear medicine departments under strict radioprotection protocols.

More recently, several healthcare institutions in France have introduced systematic clinical pharmacy activities for all patients treated with TRT, allowing for pharmaceutical validation of patient care. These activities may include:

A medication reconciliation (MR): a comprehensive list of all current and planned medications, gathered from at least three sources (e.g., prescriptions, general practitioner, medical records, and a pharmacist-led interview to gather additional details);

A basic prescription review without medication history collection;

Medication reconciliation at hospital admission or discharge.

These activities, carried out by the radiopharmacist, aim to lead to a pharmaceutical intervention (PI)-a proposal to modify a medical prescription in response to a detected medication-related issue.

This project aims to evaluate the impact of radiopharmacy activities, particularly medication reconciliation and pharmacist-patient interviews, in securing the care pathway for patients undergoing TRT. A key component of this work is the creation of a national collaborative database, in partnership with the French Society of Radiopharmacy (SOFRA). This database will also document the range of clinical radiopharmacy activities implemented across different institutions, their feasibility, the pharmaceutical interventions made, and their contributions to patient monitoring and safety.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients treated in nuclear medicine with pharmaceutical validation for a first Targeted Radionuclide Therapy (TRT) will be included in the database.
* All patients for whom a pharmaceutical intervention (PI) has been made, whether for a first or subsequent TRT.

Exclusion Criteria:

* Minor patient
* Patient without a pharmaceutical intervention for a treatment other than the first TRT course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient managed in nuclear medicine for Targeted Radionuclide Therapy (TRT) and for whom pharmaceutical validation was performed by a radiopharmacist.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the contribution of conducting a medication reconciliation to improve the safety of the care pathway for patients receiving their first Targeted Radiotherapy (initial course), compared to care without medication reconciliation | The pharmaceutical intervention will be measured at the time of interview with the patient in the group medication reconciliation AND before RIV treatment or treatment pharmaceutic order in the group solely on the patient's medical and laboratory data
  Comparison of patient care pathway safety, as measured by the rate of pharmaceutical interventions (i.e., standardized prescription modification proposals made by the radiopharmacist), in patients receiving their first Targeted Radiotherapy (TRT), following pharmaceutical validation including a medication reconciliation, versus validation based solely on the patient's medical and laboratory data.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hospices Civils de Lyon, Bron
  - CGFL Dijon, Dijon
  - Centre Hospitalier Universitaire de Lille, Lille